CLINICAL TRIAL: NCT03504969
Title: Assiut University,Faculty of Medicine
Brief Title: Perinatal Outcomes in Umbilical Cord Entanglement
Acronym: AssiutU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Gamal, Principal Investigator, Assiut University
Other Study IDs: Assiut71515
Record Dates: First submitted 2018-03-28; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Umbilical Cord; Complications, Affecting Fetus
Keywords: umbilical cord

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Umbilical Cord Entanglement and Perinatal Outcomes.

DETAILED DESCRIPTION:
Umbilical Cord Entanglement and Perinatal Outcomes neonatal outcomes and the effect on mode of delivery

ELIGIBILITY:
Inclusion Criteria:

* all vaginal deliveries with or without Umbilical Cord Entanglement

Exclusion Criteria:

* multible pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: women in active vaginal delivery
Sampling Method: Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
perinatal outcomes | one year
  number of neonates with bad Apgar score

SECONDARY OUTCOMES:
delivery outcome | one year
  number of vaginal deliveries switch to S.C